CLINICAL TRIAL: NCT06591793
Title: A Phase 1/2 Multicenter, Open-label, Dose Escalation, Safety and Efficacy Study of Subretinal Administration of Dual AAV8.MYO7A, AAVB-081 in Subjects With Usher Syndrome Type IB (USH1B) Retinitis Pigmentosa
Brief Title: Study of Subretinally Injected AAVB-081 in Patients With Usher Syndrome Type IB (USH1B) Retinitis Pigmentosa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AAVantgarde Bio Srl (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 081-101
Record Dates: First submitted 2024-08-16; First posted 2024-09-19 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Usher Syndrome, Type 1B
Keywords: Usher Syndrome; MYO7A; USH1B; Retinitis Pigmentosa
MeSH Terms: conditions — Usher syndrome, type 1B; Usher Syndromes; Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): AAVB-081 dose level 1
  Interventions: Biological: AAVB-081
- Cohort 2 (Experimental): AAVB-081 dose level 2
  Interventions: Biological: AAVB-081
- Cohort 3 (Experimental): AAVB-081 dose level 3
  Interventions: Biological: AAVB-081

INTERVENTIONS:
Biological: AAVB-081 — Single subretinal administration

SUMMARY:
The purpose of the 081-101 study is to evaluate the safety and tolerability of a single subretinal injection of AAVB-081 in USH1B patients with retinitis pigmentosa due to a mutation in the MYO7A gene. The study will also assess the initial efficacy following AAVB-081 administration.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of USB1B due to MYO7A mutation
* Willingness to adhere to protocol per informed consent

Exclusion Criteria:

* Unwillingness to meet the requirements of the study
* Participation in a clinical study with an Investigation Product in the past 6 months
* Previous participation in another Gene Therapy trial
* Any condition that would preclude subretinal surgery
* Complicating ocular and/or systemic diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
To measure the number and severity of treatment related adverse events following treatment with AAVB-081 | 61 months

SECONDARY OUTCOMES:
Change from baseline in microperimetry following treatment with AAVB-081 | 61 months
Change from baseline in static perimetry following treatment with AAVB-081 | 61 months

CONTACTS AND LOCATIONS:
Locations (3):
- University of Campania Luigi Vanvitelli, Naples, Italy
- United Kingdom (2):
  - Moorfields Eye Hospital, London
  - Retina Clinic London, London

IPD SHARING:
Plan to Share IPD: No